CLINICAL TRIAL: NCT03721055
Title: 18F-(2S,4R)4-Glutamine PET/CT in Imaging Patients With Malignant Tumor
Brief Title: Fluoroglutamine PET/CT in Imaging Patients With Malignant Tumor
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Xinhua Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: XHEC-C-2017-029-2
Record Dates: First submitted 2018-10-24; First posted 2018-10-26 (Actual); Last update posted 2019-09-06 (Actual); Status verified 2019-08

CONDITIONS: Cancer; Metastatic Cancer; Metastatic Brain Cancer
MeSH Terms: conditions — Neoplasms; Neoplasm Metastasis; Brain Neoplasms | interventions — 4-fluoroglutamine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 4-[18F]Fluoroglutamine (Experimental): Patients undergo 18F-FDG PET/CT scan first. Within 7 working days, patients receive 4-[18F]Fluoroglutamine IV and 60 minutes after injection, undergo 4-[18F]Fluoroglutamine PET/CT before the start of therapy.
  Interventions: Radiation: 18F-(2S,4R)4-fluoroglutamine

INTERVENTIONS:
Radiation: 18F-(2S,4R)4-fluoroglutamine — Undergo 18F-(2S,4R)4-fluoroglutamine PET/CT

SUMMARY:
This clinical trial studies positron emission tomography (PET) imaging utilizing 18F-(2S,4R)4-fluoroglutamine, a glutamic acid derivative, to image patients with malignant tumor. [18F]Fluoroglutamine PET may provide additional information that help diagnose and stage cancer patients.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18-79;
* The patient must be able to give informed consent;
* Patients can finish PET/CT scan without tranquilizers;
* Patients with pathology-proven cancer or a tumor highly suspected to be malignant ;
* Lesions can be measured and assessed at the RECIST 1.1 standard;
* No chemotherapy, radiotherapy or immune/biologic therapy,or biopsy were allowed between the 18F-FDG and the 4-[18F]Fluoroglutamine PET/CT.

Exclusion Criteria:

* Pregnant or lactating patients;
* Inability or refusal to have at least one peripheral intravenous line for intravenous access;
* From assays obtained <2 weeks prior to study enrollment（ULN：the upper limit of normal value ）:Bilirubin>1.5*ULN,AST/ALT >2.5 * ULN, Albumin< 3 g/dl, GGT > 2.5 x ULN if ALP> 2.5 x ULN, Creatinine>1.5*ULN or creatinine clearance <60ml/min；
* Patients with a history of allergic reaction to this drugs or its analogues；
* patients with poor compliance;
* Acute major illness

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2017-08-21 (Actual); Primary Completion 2019-12-31 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
Diagnosing and Staging ability of 4-[18F]Fluoroglutamine PET/CT in malignant cancer | up to three years
  Sensitivity, specificity, diagnostic accuracy of 4-[18F]Fluoroglutamine and 18F-FDG PET/CT will be compared using paired t-test or Krusal-Wallis test.

SECONDARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events | up to 30 days after the F-Gln imaging
  The evaluation of the Incidence of Treatment-Emergent Adverse Events starts from the day of F-Gln examination until 30 days later; Treatment-Emergent Adverse Events are evaluated according to version 4.03 CTC-AE criteria.
ASCT2 expression levels in tissue samples | up to three years
  Wilcoxon rank-sum or Kruskal-Wallis tests will be applied for the group comparisons of IHC staining(ASCT2)
The correlation between 18F-(2S,4R)4- glutamine PET/CT imaging and prognosis in malignant tumors | up to three years
  Evaluating the prognostic value of metabolic parameters and clinical indexes by using log-rank tests on univariate analysis and COX proportional hazards regression tests

CONTACTS AND LOCATIONS:
Locations (1):
- Xinhua Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided